CLINICAL TRIAL: NCT00817037
Title: The Effect of Sitaxsentan Once Daily Dosing on Proteinuria, 24-hour Systemic Blood Pressure, and Arterial Stiffness in Subjects With Chronic Kidney Disease
Brief Title: Sitaxsentan in Proteinuric Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Encysive Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007/W/CRC/02; CTA# 2006-002004-33; 06/MRE10/69
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Chronic Kidney Disease; Proteinuria; Blood Pressure
Keywords: Chronic kidney disease; Proteinuria; Blood pressure; Arterial stiffness; Endothelin antagonist; Sitaxsentan
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria | interventions — sitaxsentan; Nifedipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sitaxsentan (Experimental): Once daily oral sitaxsentan 100mg given over a period of 6 weeks.
  24hr proteinuria, 24hr blood pressure and arterial stiffness measured at day 1, week 3 and week 6 of treatment
  Interventions: Drug: Sitaxsentan
- Placebo (Placebo Comparator): Once daily oral placebo tablet given over a period of 6 weeks.
  24hr proteinuria, 24hr blood pressure and arterial stiffness measured at day 1, week 3 and week 6 of treatment
  Interventions: Drug: Placebo tablet
- Nifedipine (Active Comparator): Open labeled active comparator
  Once daily oral nifedipine 30mg given over a period of 6 weeks.
  24hr proteinuria, 24hr blood pressure and arterial stiffness measured at day 1, week 3 and week 6 of treatment
  Interventions: Drug: Nifedipine

INTERVENTIONS:
Drug: Sitaxsentan — Sitaxsentan 100mg once daily oral dosing for 6 weeks
  Other Names: Thelin
  Arms: Sitaxsentan
Drug: Nifedipine — Nifedipine 30mg once daily oral dosing for 6 weeks
  Other Names: Adalat LA
  Arms: Nifedipine
Drug: Placebo tablet — Placebo tablet once daily oral dosing for 6 weeks
  Arms: Placebo

SUMMARY:
Patients with chronic kidney disease (CKD) have higher blood pressures than the general population. They also tend to have protein leaking into the urine (proteinuria). CKD, high blood pressure and proteinuria independently and together increase the risk of developing atherosclerosis (hardening) of the arteries that leads to diseases such as heart attack and stroke. Although there are a number of drugs available that lower blood pressure, these are not always fully effective. Furthermore, there are even fewer drugs that simultaneously lower blood pressure, reduce proteinuria, and slow down kidney damage in CKD.

Recent research has shown that drugs like sitaxsentan not only lower blood pressure but also reduce proteinuria and potentially slow down the progression of CKD [1,2]. Before sitaxsentan can become freely available to individuals with CKD it is important to look at the effects this drug could have on proteinuria and blood pressure.

1. Goddard J, Johnston NR, Hand MF, et al. Endothelin-A receptor antagonism reduces blood pressure and increases renal blood flow in hypertensive patients with chronic renal failure: a comparison of selective and combined endothelin receptor blockade. Circulation 2004;109:1186-1193.
2. Krum H, Viskoper RJ, Lacourciere Y et al. The effect of an endothelin receptor antagonist, bosentan, on blood pressure in patients with essential hypertension. New Engl J Med 1998;338:784-790.

ELIGIBILITY:
Inclusion Criteria:

1. Has Stage 1-5 chronic kidney disease (CKD) as defined by the Kidney Disease Outcomes Quality Initiative (using the Cockcroft and Gault equation for calculation of glomerular filtration rate) with proteinuria, including any of the following aetiologies: immunoglobulin A (IgA) nephropathy, polycystic kidney disease (PCKD), congenital abnormalities, reflux nephropathy, focal segmental glomerulosclerosis, minimal change nephropathy, and membranous nephropathy.
2. Is between 18 and 70 years of age, inclusive.
3. Has a body mass index (BMI) between 18 and 35 kg/m2, inclusive.
4. Is willing and able to adhere to the protocol requirements.
5. Provides written informed consent before any study procedure is performed.

Exclusion Criteria:

1. Requires peritoneal dialysis or haemodialysis.
2. Has kidney disease due to diabetes mellitus, vasculitis, systemic lupus erythematosus, or known renovascular disease; antiglomerular basement membrane disease; or is on immunosuppressive medication.
3. Has a serum albumin in the nephrotic range (< 30 g/L) during Screening.
4. Has a sustained sitting systolic blood pressure (BP) > 160 mmHg or sustained sitting diastolic BP > 100 mmHg during Screening.
5. Has postural hypotension during Screening, which is defined as a decrease in systolic BP ≥ 20 mmHg and/or a decrease in diastolic BP ≥ 10 mmHg, comparing sitting and standing measurements.
6. Has a history and/or evidence of ischaemic heart disease.
7. Has or had a malignancy, with the exception of adequately-treated basal cell or squamous cell carcinoma of the skin, that required significant medical intervention within the past 3 months and/or is likely to result in death within the next 2 years.
8. Has a history of allergies or hypersensitivity to sitaxsentan or nifedipine or the excipients of either drug.
9. Has a clinically significant psychiatric, addictive, neurological disease or any other condition that, in the Investigator's opinion, would compromise his/her ability to give informed consent, participate fully in this study, prevent adherence to the requirements of the study protocol, or would compromise the interpretation of the data obtained from this study.
10. Uses a prohibited medication or plans to use a prohibited medication during the study.

    * Prohibited medications include cyclosporine A, alternative endothelin (ET) receptor antagonists, phosphodiesterase inhibitors, and/or vitamin K antagonists (e.g., warfarin). The intermittent use of phosphodiesterase inhibitors (e.g., sildenafil) "as needed" for erectile dysfunction is acceptable, however, as long as the subject is not dosed within 24 hours of an efficacy assessment.
11. Received treatment with an investigational drug or device within 30 days prior to study entry.
12. Has a history of organ transplantation.
13. Has atrial fibrillation requiring anticoagulation or a history (in the preceding 6 months) of any intermittent cardiac dysrhythmia that may require anticoagulation therapy.
14. Has an alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) level > 1.5 × the upper limit of the normal range (ULN) at Screening and/or serum total bilirubin > ULN.
15. Has a haemoglobin concentration < 8.0 mg/dL at Screening.
16. Has positive serological results for hepatitis B and/or hepatitis C.
17. Is a woman of childbearing potential who is unwilling to use 2 forms of contraceptive therapy, including at least 1 barrier method, throughout the study. (Women who are surgically sterile or who are post-menopausal for at least 2 years are not considered to be of childbearing potential.)
18. Is pregnant, lactating, or breastfeeding.
19. Has, in the opinion of the Investigator, a dependence on alcohol.
20. Has, in the opinion of the Investigator, a dependence on illicit drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-07-14 (Actual); Primary Completion 2009-07-07 (Actual); Study Completion 2009-07-07 (Actual)

PRIMARY OUTCOMES:
The principal objective of this study is to evaluate whether sitaxsentan reduces proteinuria in people with chronic kidney disease. | 6 Weeks

SECONDARY OUTCOMES:
Secondary objective of this study is to evaluate whether sitaxsentan reduces systemic blood pressure in people with chronic kidney disease. | 6 weeks
Secondary objective is to determine whether sitaxsentan improves indices of arterial stiffness in people with chronic kidney disease | 6 weeks
Secondary objectives is to determine the safety of sitaxsentan in chronic kidney disease | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Webb, MD DSc FRCP FRSE FMedSci, Study Director — University of Edinburgh; Neeraj Dhaun, MBChB, Principal Investigator — University of Edinburgh
Locations (1):
- Clinical Research Centre, Western General Hospital, Edinburgh, Scotland, United Kingdom